CLINICAL TRIAL: NCT02549833
Title: Pilot Randomized Neo-adjuvant Evaluation of Poly-ICLC-Assisted Tumor Lysate Vaccines in Adult Patients With WHO Grade II Glioma
Brief Title: Neo-adjuvant Evaluation of Glioma Lysate Vaccines in WHO Grade II Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennie Taylor (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Jennie Taylor, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-17692; 15103 (Other: University of California, San Francisco); NCI-2017-01683 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-08-20; First posted 2015-09-15 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Oligodendroglioma; Astrocytoma, Grade II; Glioma, Astrocytic; Glioma; Malignant Glioma; Oligoastrocytoma, Mixed
Keywords: low-grade glioma; WHO grade II; vaccine; immunotherapy; glioma
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma; Glioma; Lymphoma, Follicular | interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaccines before and after surgery (Experimental): GBM6-AD lysate protein 1 mg and poly-ICLC 1.4 mg administered as one formulation every week leading up to standard-of-care surgery to remove the WHO grade II glioma (Days -23±2, -16±2, -9±2 and 24-48 hours prior to scheduled surgery), every 3 weeks after surgery (Weeks A1, A4, A7, A10, A13, A16; defining Week A1 as the first post-surgery vaccine), and two booster vaccines (Weeks A32 and A48).
  Interventions: Biological: GBM6-AD and poly-ICLC before and after surgery
- Vaccines after surgery only (Active Comparator): GBM6-AD lysate protein 1 mg and poly-ICLC 1.4 mg administered as one formulation every 3 weeks after standard-of-care surgery to remove the WHO grade II glioma only (Weeks A1, A4, A7, A10, A13, A16; defining Week A1 as the first post-surgery vaccine) and two booster vaccines (Weeks A32 and A48). Patients will not receive vaccines before surgery.
  Interventions: Biological: GBM6-AD and poly-ICLC after surgery only

INTERVENTIONS:
Biological: GBM6-AD and poly-ICLC before and after surgery — Subcutaneous vaccination with GBM6-AD lysate protein and poly-ICLC combination
  Arms: Vaccines before and after surgery
Biological: GBM6-AD and poly-ICLC after surgery only — Subcutaneous vaccination with GBM6-AD lysate protein and poly-ICLC combination
  Arms: Vaccines after surgery only

SUMMARY:
This is a pilot neoadjuvant vaccine study in adults with WHO grade II glioma, for which surgical resection of the tumor is clinically indicated. Co-primary objectives are to determine: 1) the safety and feasibility of the neoadjuvant approach; and 2) whether the regimen increases the level of type-1 chemokine CXCL10 and vaccine-specific (i.e., reactive to GBM6-AD) CD8+ T-cells in tumor-infiltrating leukocytes (TILs) in the surgically resected glioma.

DETAILED DESCRIPTION:
Low-grade gliomas (LGG), the most common of which are pilocytic astrocytomas, diffuse astrocytomas, oligodendrogliomas, and mixed oligo-astrocytomas are a diverse family of central nervous system (CNS) neoplasms that occur in children and adults. Based on data from the American Cancer Society and Central Brain Tumor Registry of the United States (CBRTUS), approximately 1800 LGG were diagnosed in 2006, thus representing approximately 10% of newly diagnosed primary brain tumors in the United States. Pilocytic astrocytomas (WHO grade I) are the most common brain tumor in children 5 to 19 years of age3. Diffuse astrocytomas, oligodendrogliomas, and oligoastrocytomas are all considered WHO grade II low grade gliomas (LGG) and are more common in adults. Pilocytic astrocytomas are generally well circumscribed histologically and radiographically and amenable to cure with gross total resection. In contrast, the diffuse astrocytomas, oligodendrogliomas, and oligoastrocytomas are more infiltrative and less amenable to complete resection. From a molecular genetics standpoint, the most common alterations in LGG are Isocitrate dehydrogenase 1 (IDH1) mutations and mutations in the tumor suppressor gene TP53, located on chromosome 17, the gene product of which is a multifunctional protein involved in the regulation of cell growth, cell death (apoptosis), and transcription. Additionally, several molecular factors are of favorable prognostic significance, particularly the presence of 1p/19q co-deletion and IDH1 mutations.

WHO grade II LGGs are at extremely high risk to undergo malignant transformation into more aggressive and lethal WHO grade III or IV high-grade glioma (HGG). Even with a combination of available therapeutic modalities (i.e., surgery, radiation therapy [RT], chemotherapy), the invasive growth and resistance to therapy exhibited by these tumors results in recurrence and death in most patients. Although postoperative RT in LGG significantly improves 5-year progression-free survival (PFS), it does not prolong overall survival (OS) compared with delayed RT given at the time of progression. Early results from a randomized trial of radiation therapy plus procarbazine, lomustine, and vincristine (PCV) chemotherapy for supratentorial adult LGG (RTOG 9802) demonstrated improved PFS in patients receiving PCV plus RT compared RT alone. Nonetheless, PCV is considerably toxic and currently not widely used for management of glioma patients. Although chemotherapy with temozolomide (TMZ) is currently being investigated in LGG patients, it is unknown whether it confers improves OS in these patients. Further, our recent study has indicated that 6 of 10 LGG cases treated with TMZ progressed to HGG with markedly increased exome mutations and, more worrisome, driver mutations in the RB and protein kinase B (AKT)-mechanistic target of rapamycin (mTOR) pathways, with predominant C>T/G>A transitions at CpC and CpT dinucleotides, strongly suggesting a signature of TMZ-induced mutagenesis; this study also showed that in 43% of cases, at least half of the mutations in the initial tumor were undetected at recurrence. These data suggests the possibility that treatment of LGG patients with TMZ may enhance oncogenic mutations and genetic elusiveness of LGG, therefore calling for development of safer and effective therapeutic modalities such as vaccines.

Taken together, LGG are considered a premalignant condition for HGG, such that novel interventions to prevent malignant transformation need to be evaluated in patients with LGG. Immunotherapeutic modalities, such as vaccines, may offer a safe and effective option for these patients due to the slower growth rate of LGG (in contrast with HGG), which should allow sufficient time for multiple immunizations and hence high levels of anti-glioma immunity. Because patients with LGGs are generally not as immuno-compromised as patients with HGG, they may also exhibit greater immunological response to and benefit from the vaccines. Further, the generally mild toxicity of vaccines may improve quality of life compared with chemotherapy or RT.

ELIGIBILITY:
Inclusion Criteria:

* Pathological criteria - Patients must have newly diagnosed or recurrent WHO grade II glioma (defined as an astrocytoma, oligodendroglioma, or oligoastrocytoma) that is to be histologically confirmed by clinically indicated resection. If patients have already undergone biopsy and have pathological diagnosis of WHO grade II glioma, pathology must be reviewed and confirmed at University of California, San Francisco (UCSF).
* Before enrollment, patients must show supratentorial, non-enhancing T2-FLAIR lesions that need to be surgically resected and are likely WHO grade II glioma. Surgical resection of at least 500 mg tumor tissue to ensure adequate evaluation of the study endpoints.
* Prior radiation therapy (RT) after the initial diagnosis will be allowed. Patients with prior RT must be at least 6 months from the completion of RT (or radiosurgery)
* Prior chemotherapy or molecularly targeted therapy will be allowed. Patients with prior chemotherapy must be at least 6 months from the last dose of chemotherapy or molecularly targeted therapy
* Patients must be ≥ 18 years old
* Patients must have a Karnofsky performance status ≥ 70%
* Patients must be off corticosteroid for at least for 2 weeks before the first neoadjuvant vaccine and for at least 2 weeks prior to the first adjuvant vaccine
* Adequate organ function within 14 days of study registration including:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1.0 x 10^9/L; absolute lymphocyte count (ALC) ≥0.5 x 10^9/L; platelets ≥100 x 10^9/L; hemoglobin ≥8 g/dL;
  * Hepatic: - Total bilirubin ≤1.5 x upper limit of normal (ULN) and serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase (ALT)) ≤ 2.5 x upper limit of normal (ULN), and
  * Renal: Normal serum creatinine or creatinine clearance ≥60 ml/min/1.73 m^2
* Must be free of systemic infection. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.
* Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device (IUD), surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of the vaccination period. Sexually active males must agree to use barrier contraceptive for the duration of the vaccination period.

Exclusion Criteria:

* History of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, transplant immunosuppression)
* History or clinical suspicion of neurofibromatosis
* Any isolated laboratory abnormality suggestive of a serious autoimmune disease (e.g. hypothyroidism)
* Any conditions that could potentially alter immune function (AIDS, multiple sclerosis, uncontrolled diabetes, renal failure)
* Receiving ongoing treatment with immunosuppressive drugs
* Currently receiving any investigational agents or registration on another therapy based trial
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Regimen Limiting Toxicity (RLT) | until disease progression, start of a new therapy, or for a maximum of 18 months from study registration (whichever occurs earlier)
  Delay of the scheduled surgery for longer than 2 weeks due to toxicity of the neoadjuvant treatment will also be considered RLT and reported for each arm will be tabulated with 95% exact (ClopperPearson) confidence intervals
Measurement of vaccine-induced immune response in the resected tumor | At time of surgery (as clinically indicated)
  Evaluate whether surgically resected tumors from Arm 1 (the neoadjuvant arm) patients demonstrate significantly higher levels of CD8+ T-cell infiltration and CXCL10 expression compared with those resected from Arm 2 (control) patients The mean CD8+ T-cells in TILs and CXCL10 expression will be compared between arms by means of a two-sample Student's t test. If the t test assumptions are not met and the data cannot be transformed in such a way that the assumptions are met, a Wilcoxon Rank Sum test will be used

SECONDARY OUTCOMES:
Response rate of CD4+ and CD8+ T-cell responses against the GM6-AD lysate in pre- and post-vaccine peripheral blood mononuclear cell (PBMC) using IFN-γ-ELISPOT | at Baseline, At time of surgery (as clinically indicated), Weeks 1, 10 and 16 post-surgery
  To describe the response rate and magnitude of CD4+ and CD8+ T-cell responses against the GBM6-AD lysate in pre- and postvaccine PBMC using interferon (IFN)-γ-ELISPOT. Further, we will determine whether T-cell clonotypes changes in PBMC during the course of the vaccines. We will also determine whether T-cell clonotypes that increased in post-vaccine PBMC are found in tumor infiltrating lymphocytes (TILs).
Magnitude of response of CD4+ and CD8+ T-cell responses against the GM6-AD lysate in pre- and post-vaccine PBMC using IFN-γ-ELISPOT | at Baseline, At time of surgery (as clinically indicated), Weeks 1, 10 and 16 post-surgery
  To describe the response rate and magnitude of CD4+ and CD8+ T-cell responses against the GBM6-AD lysate in pre- and postvaccine PBMC using interferon (IFN)-γ-ELISPOT. Further, we will determine whether T-cell clonotypes changes in PBMC during the course of the vaccines. We will also determine whether T-cell clonotypes that increased in post-vaccine PBMC are found in tumor infiltrating lymphocytes (TILs).
Tumor tissue expression of glioma-associated antigens (GAAs) and antigen-presentation machinery (APM) molecules | At the time of clinically indicated surgical resection of the tumor
  To describe tumor tissue expression of glioma-associated antigens (GAAs) and antigen-presentation machinery (APM) molecules. We will evaluate whether there are changes in GAA and APM expression status over the course
Overall survival (OS) | Minimum of 2 years
  OS is defined as the duration of time from start of treatment to death. All patients will be followed for a minimum of 2 years
Objective response rate (ORR) | Minimum of 2 years
  objective response rate (ORR) will be tabulated by response according to low-grade gliomas (LGG) Response Assessment in Neuro-Oncology (RANO)
Progression-free survival (PFS) | Minimum of 2 years
  PFS is defined as the duration of time from start of treatment to time of progression. All patients will be followed for a minimum of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Taylor, MD, Principal Investigator — University of California, San Francisco; Hideho Okada, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogino H, Taylor JW, Nejo T, Gibson D, Watchmaker PB, Okada K, Saijo A, Tedesco MR, Shai A, Wong CM, Rabbitt JE, Olin MR, Moertel CL, Nishioka Y, Salazar AM, Molinaro AM, Phillips JJ, Butowski NA, Clarke JL, Oberheim Bush NA, Hervey-Jumper SL, Theodosopoulos P, Chang SM, Berger MS, Okada H. Randomized trial of neoadjuvant vaccination with tumor-cell lysate induces T cell response in low-grade gliomas. J Clin Invest. 2022 Feb 1;132(3):e151239. doi: 10.1172/JCI151239. PMID 34882581